CLINICAL TRIAL: NCT03297398
Title: A Randomized, Double-blind, Placebo-controlled Dose-ranging Study of OPK-88004 Once-a-day Dosing for 16 Weeks in Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Effects and Safety of OPK-88004 Doses in Men With Signs and Symptoms of Benign Prostatic Hyperplasia (BPH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study terminated by sponsor decision
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAR-202
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Other (Placebo Comparator): Placebo Group
  Interventions: Other: Placebo
- Drug Group 1 (Experimental): 15mg, OPK-88004
  Interventions: Drug: Group-1 (15mg, OPK-88004)
- Drug Group 2 (Experimental): 25,mg OPK-88004
  Interventions: Drug: Group-2 (25 mg,OPK-88004)

INTERVENTIONS:
Drug: Group-1 (15mg, OPK-88004) — 15mg, OPK-88004
  Other Names: Selective Androgen Receptor Modulator
  Arms: Drug Group 1
Drug: Group-2 (25 mg,OPK-88004) — 25 mg,OPK-88004
  Other Names: Selective Androgen Receptor Modulator
  Arms: Drug Group 2
Other: Placebo — Placebo
  Other Names: Inactive
  Arms: Other

SUMMARY:
This study will evaluate the safety and effectiveness of different doses of OPK-88004 compared to placebo on serum PSA compared to placebo in men with benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
Study SAR-202 is a phase 2 multicenter, placebo-controlled, double-blind trial to evaluate the effect of OPK-88004 doses (OPK-88004 15 mg, or OPK-88004 25 mg) on serum PSA compared to placebo in men with BPH. Approximately 115 men with BPH will be enrolled in the study, randomized 1:1:1 across three arms (placebo, OPK-88004 15 mg, or OPK-88004 25 mg). The trial will be conducted at approximately up to 35 sites within the US.

The study duration for individual subjects will be up to 24 weeks and will include three phases:

* a screening period (up to 4 weeks, including 1-week washout if required),
* a treatment period (16 weeks), and
* a follow-up period (4 weeks) Subjects will be randomized and receive their first dose of study drug at visit 2. They will begin the once daily oral dosing regimen and return every 4 weeks to the study site during the 16-week treatment period. Assessments during the study period will include vital signs, laboratory testing, weight, adverse events (AEs), concomitant drugs, and study drug compliance. Efficacy assessments will include serum PSA, LBM and fat mass by DXA scans, uroflowmetry parameters, PVR (by ultrasound), and assessment of symptoms by IPSS.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible if they meet the following criteria:

1. Present with BPH-LUTS based on disease diagnostic criteria at visit 1
2. Are men aged 45 years or older at visit 1
3. Have prostate volume >40 cm3 and <80 cm3 assessed by TRUS at visit 1
4. Have a PSA >1.5 and <10.0 ng/mL at visit 1. This PSA blood draw must be performed at least 1 week after any digital rectal exam (DRE) and/or transrectal ultrasound (TRUS) procedures
5. Subjects with a PSA ≥4.0 and <10.0 ng/mL must have documentation of a negative histologic biopsy of carcinoma of the prostate within 12 months of screening (visit 1). For subjects aged ≤80 years and who have not undergone any invasive urological procedure within 6 months, if biopsy has not been performed, then 4Kscore Test value must be <7.5% at visit 1
6. Have laboratory tests within normal limits (with the exception of total serum or free testosterone). If laboratory test results are outside normal limits they are determined to be not clinically significant at visit 1
7. Have not received prior treatment with 5-ARIs (finasteride, dutasteride) within the past one year for any indication
8. Have not received herbal BPH preparations within 1 week of visit 1. If the subject is currently on such treatment, a 1-week washout period will be required
9. Agree not to use 5-ARIs, herbal or experimental treatments for BPH, at any time during the study. Subjects on daily PDE5i's, alpha-blockers or anticholinergic medications for BPH should remain on a stable dose during the study, unless a change in dose is medically warranted. Occasional-use PDE5i's for ED are permitted at a stable dose and frequency, however should not be taken within 72 hours prior to a study visit
10. Agree to use an acceptable method of birth control during the study and for 60 days after the last dose of IP, unless the female partner is postmenopausal. Postmenopausal is defined as a female >50 years of age and 12 months of amenorrhea, or surgically postmenopausal
11. Are reliable and willing to make themselves available for the duration of the study, and who will comply with the required study and dosing visits and abide by the Clinical Research Site policy and procedure and study restrictions
12. Have given written informed consent

Exclusion Criteria

Patients will be excluded from study enrollment if they meet any of the following criteria at visit 1:

1. History of any of the following pelvic conditions:

   * radical prostatectomy, pelvic surgery for removal of malignancy, or bowel resection
   * pelvic radiotherapy
   * any pelvic surgical procedure on the urinary tract, including transurethral resection of the prostate (TURP), penile implant surgery
   * lower urinary tract malignancy or trauma
   * pelvic surgery or any other pelvic procedure less than 6 months prior to visit 1
2. Lower urinary tract instrumentation (including prostate biopsy) within 6 weeks prior to screening PSA blood draw
3. History of urinary retention or lower urinary tract (bladder) stones within 1 month of visit 1
4. Minimally invasive procedures for BPH, such as prostatic stent, high intensity focused ultrasound (HIFU), holmium laser enucleation of prostate (HoLEP), interstitial laser coagulation (ILC), transurethral electroevaporation of the prostate (TUVP), transurethral microwave thermotherapy (TUMT), transurethral needle ablation (TUNA), photoselective vaporization (PVP), UroLift, within 6 weeks
5. Clinical evidence of urinary tract infection or urinary tract inflammation (including prostatitis)
6. Intravesical obstruction (eg, intravesical median lobe of the prostate)
7. Current neurologic disease or condition associated with neurogenic bladder (eg, Parkinson's disease, multiple sclerosis)
8. History of significant renal insufficiency, defined as receiving renal dialysis or having an estimated creatinine clearance <45 mL/min
9. Active hepatobiliary disease or serologic evidence of active hepatitis A, B, C, hepatitis E or HIV
10. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 2X the upper limit of normal (ULN)
11. Glycosylated hemoglobin (HbA1c) >9%
12. Hematocrit ≥50%
13. HDL-C <35 mg/dL and LDL-C >130 mg/dL
14. QTcB interval >450 msec. For heart rates over 75, the ECG may be repeated after 5 minutes of resting quietly
15. Abnormality in ECG (eg, left bundle branch block, complete right bundle branch block, or delayed intraventricular conduction with a QRS interval >120 msec) that in the opinion of the investigator places the subject at an unacceptable risk for study participation, or subject has implanted pacemaker
16. History of any of the following cardiac/coronary conditions within 90 days:

    * history of myocardial infarction or coronary artery bypass graft
    * percutaneous coronary intervention
    * stroke
17. Any evidence of heart disease (NYHA ≥Class II, Appendix 4) within 6 months, or are receiving treatment for congestive heart failure (CHF)
18. Any supraventricular or ventricular arrhythmia with uncontrolled ventricular response (mean heart rate >100 bpm) at rest despite medical therapy
19. Systolic blood pressure >160 or <90 mm Hg or diastolic blood pressure >100 or <50 mm Hg as determined by a sitting measurement (if stress is suspected, retest up to two times under basal conditions), or malignant hypertension
20. Have a history or presence of prostatic carcinoma, as well as any conditions that may be exacerbated by androgenic medications such as (but not limited to) epilepsy, seizures, convulsions, migraine or polycythemia
21. History of cancer within the previous 5 years, except for excised superﬁcial lesions (such as basal cell carcinoma and squamous cell carcinoma of the skin)
22. History of drug, alcohol, or substance abuse within 6 months
23. Have an alcohol intake of ≥3 units/day or ≥14 units/week during the study (1 unit = 12 ounces of beer, 5 ounces of wine, 1.5 ounces of distilled spirits)
24. Any condition that would interfere with subject's ability to provide informed consent or comply with study instructions, would impair ability to perform the study assessments, or would place subject at increased risk, or might confound the interpretation of the study results
25. Current treatment with androgens, antiandrogens, estrogens, or anabolic steroids within the prior 1 month. Any prior or current treatment with LHRH agonists/antagonists
26. Current treatment with potent CYP3A4 inhibitors such as itraconazole or ritonavir
27. Have taken prescription or over-the-counter medications to promote weight loss within the prior 3 months
28. Any prior use of OPK-88004 Allergic to any component of OPK-88004

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Militza Vera De Alba, MD, Study Director — Dr.
Locations (15):
- United States (15):
  - Pinnacle Research Group, Anniston, Alabama
  - Clinical Trials Research, Lincoln, California
  - Northern California Research, Sacramento, California
  - Bayview Research Group, LLC - Valley Village, Valley Village, California
  - South Florida Medical Research, Aventura, Florida
  - APF Research, LLC, Miami, Florida
  - Meridien Research - Brooksville, Spring Hill, Florida
  - Florida Urology Partners, Tampa, Florida
  - Advanced Clinical Research - Boise, Meridian, Idaho
  - Regional Urology, Shreveport, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - Volunteer Research Group and New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo Group
  Placebo: Placebo
- OPK-88004 15 mg: 15mg, OPK-88004
  Group-1 (15mg, OPK-88004): 15mg, OPK-88004
- OPK-88004 25 mg: 25mg, OPK-88004
  Group-2 (25 mg,OPK-88004): 25 mg,OPK-88004
Period: Overall Study
Arm/Group | Placebo | OPK-88004 15 mg | OPK-88004 25 mg
Started | 36 | 40 | 38
Completed | 28 | 23 | 23
Not Completed | 8 | 17 | 15
Not completed — Sponsor's decision | 6 | 9 | 7
Not completed — Adverse Event | 1 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Other | Drug Group 1 | Drug Group 2 | Total
Number analyzed (Participants) | 36 | 40 | 38 | 114
Age, Continuous [Mean (Standard Deviation); unit: Year] | 64.1 (6.52) | 64.5 (5.77) | 65.3 (6.01) | 64.6 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 36 | 40 | 38 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 5 | 15
  Not Hispanic or Latino | 29 | 37 | 33 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight (kilogram) [Mean (Standard Deviation); unit: Kilogram] | 94.97 (16.937) | 95.31 (19.128) | 91.35 (13.564) | 93.88 (16.692)
Body mass index (kilogram/meter^2) [Mean (Standard Deviation); unit: Kilogram/meter^2] | 30.17 (5.114) | 30.37 (5.286) | 29.36 (3.442) | 29.97 (4.671)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PSA (%) to Week 16
Description: The trial will evaluate the effect of two doses of OPK-88004 (15 mg and 25 mg) daily for 16 weeks on serum PSA compared with placebo
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: Percentage of serum PSA change
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 36 | 38 | 35
Percentage of serum PSA change | -2.96 (5.198) | -1.48 (5.569) | -15.44 (5.509)

2. Secondary Outcome: Absolute Change in Lean Body Mass and Fat Mass From Baseline to 16 Weeks
Description: To assess the effect of OPK-88004 on body composition by DXA, specifically Lean Body Mass (LBM) and fat mass
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: gram
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 36 | 38 | 35
gram
  Change from Baseline in Lean Body Mass (g) to Week 16 | 37.8 (439.62) | 1610.3 (489.45) | 1961.6 (522.58)
  Change from Baseline in Fat Mass (g) to Week 16 | -198.2 (326.84) | -1468.7 (373.06) | -1491.3 (388.98)

3. Other Pre Specified Outcome: To Evaluate the Effect of OPK-88004 on Uroflowmetry Parameter- Peak Flow Rate (Qmax)
Description: Analysis peak flow rate of Uroflowmetry Parameters and Postvoid Residual Volume Observed Change from Baseline to Week 16
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: millilitre/second
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 33 | 29 | 28
millilitre/second | 4.26 (3.810) | 0.61 (4.072) | 1.08 (4.043)

4. Other Pre Specified Outcome: To Evaluate the Effect of OPK-88004 on Uroflowmetry Parameter- Mean Flow Rate (Qave)
Description: Analysis mean flow rate of Uroflowmetry Parameters and Postvoid Residual Volume Observed Change from Baseline to Week 16
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: millilitre/second
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 33 | 29 | 28
millilitre/second | -0.40 (0.475) | -0.30 (0.509) | 0.15 (0.505)

5. Other Pre Specified Outcome: To Evaluate the Effect of OPK-88004 on Uroflowmetry Parameter-voided Volume (Vcomp)
Description: Analysis voided of Uroflowmetry Parameters and Postvoid Residual Volume Observed Change from Baseline to Week 16
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: millilitre
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 32 | 28 | 28
millilitre | -49.12 (21.294) | -2.28 (22.501) | -29.12 (22.714)

6. Other Pre Specified Outcome: To Evaluate the Effect of OPK-88004 on Uroflowmetry Parameter- Postvoid Residual Volume (PVR)
Description: Analysis postvoid residual volume of Uroflowmetry Parameters and Postvoid Residual Volume Observed Change from Baseline to Week 16
Time Frame: 16 weeks
Measure: Least Squares Mean (Standard Error); unit: millilitre
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 32 | 28 | 29
millilitre | -0.08 (10.365) | 17.63 (11.325) | -15.19 (10.925)

7. Other Pre Specified Outcome: International Prostate Symptom Score- IPSS
Description: To evaluate the effects of OPK-88004 on the symptoms of BPH as determined by International prostate symptom score (IPSS score), Total IPSS score as measured by the sum of questions 1 through 7, the IPSS Irritative Domain (sum of questions 2, 4 and 7), and the IPSS Obstructive Domain (sum of questions 1, 3, 5 and 6)IPSS QoL question (IPSS question 8). Mild (symptoms score less than or equal to 7), moderate (symptoms score range 8-19), severe (symptom score 20-35)
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Total IPSS score
Arm/Group | Other | Drug Group 1 | Drug Group 2
Number analyzed (Participants) | 28 | 23 | 22
Total IPSS score | 14.0 (7.70) | 12.8 (6.21) | 14.2 (7.28)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Other | Drug Group 1 | Drug Group 2
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/40 | 2/38
Other Adverse Events (participants affected / at risk) | 5/36 | 25/40 | 30/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Other (N=36) | Drug Group 1 (N=40) | Drug Group 2 (N=38)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Other (N=36) | Drug Group 1 (N=40) | Drug Group 2 (N=38)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 2
Blood testosterone decreased (Investigations) | 0 | 7 | 5
Low density lipoprotein increased (Investigations) | 0 | 3 | 3
Transaminases increased (Investigations) | 1 | 2 | 3
High density lipoprotein decreased (Investigations) | 0 | 1 | 4
Prostatic specific antigen increased (Investigations) | 0 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 2
Blood testosterone free decreased (Investigations) | 0 | 1 | 3
Sperm concentration decreased (Investigations) | 0 | 1 | 3
Apolipoprotein B increased (Investigations) | 0 | 3 | 0
Blood cholesterol increased (Investigations) | 0 | 2 | 0
Blood creatine increased (Investigations) | 0 | 0 | 2
Liver function test increased (Investigations) | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Headache (Nervous system disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The obligations of non-disclosure and non-use set forth in the confidentiality is 10 years after expiration of the agreement

DOCUMENTS (2):
  • Study Protocol (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03297398/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT03297398/SAP_001.pdf